CLINICAL TRIAL: NCT04789460
Title: Relationship Between Potential Predictors and Mortality in COVID-19 Patients in Turkey: A New Prognostic Model
Brief Title: Relationship Between Potential Predictors and Mortality in COVID-19 Patients ın Turkey
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: TURKEYPROMOD
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: covid19; ldh; ferritin; mortality; d-dimer
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients in hospital: All patients aged 18 years and over, positive for SARS-CoV-2 PCR test and / or Covid-19 treatment with signs of Covid-19 disease on CT in two tertier hospital in Istanbul

SUMMARY:
In this study, the investigators planned to examine the laboratory characteristics of patients hospitalized with the diagnosis of Covid-19 and to investigate their relationship with mortality.

DETAILED DESCRIPTION:
SARS-CoV-2 infection is effective in many countries and has caused pandemics. It is observed that it affects patients in a wide spectrum in terms of their clinical features worldwide. It is known that age, gender, and comorbidity play an important role in the course of the disease. Although mortality rates vary from country to country, there is no clear information due to the fact that the pandemic has not yet ended. In this study, the investigators planned to examine the laboratory characteristics of patients hospitalized with the diagnosis of Covid-19 and to investigate their relationship with mortality in Istanbul city which is the most affected by the pandemic in Turkey

ELIGIBILITY:
Inclusion Criteria:

* All patients who are 18 years of age and older, positive for SARS-CoV-2 PCR test and / or Covid-19 disease findings on CT will be included in the study.

Exclusion Criteria:

* Patients with negative SARS-CoV-2 PCR test, pneumonia on CT but not given Covid-19 treatment by not considering Covid-19 by their doctor will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with the diagnosis of covid-19
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
mortality rate | up to 30 days
  up to 30 days after discharge

SECONDARY OUTCOMES:
need for intensive care unit rate | up to 30 days
  need for intensive care unit during hospitalization
length stay in hospital | up to 30 days
  number of length stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Han Training and Rsearch Hospital
Locations (1):
- SBU Sultan Abdulhamid Han, Istanbul, Asia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided